CLINICAL TRIAL: NCT05184894
Title: AKI in Care Transitions (ACT) Trial
Brief Title: A Study of Acute Kidney Injury in Care Transitions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Erin Barreto, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-011055; R03HS028060-01 (AHRQ)
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Patient Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AKI in Care Transitions (ACT) Group (Experimental): Subjects diagnosed with Acute Kidney Injury (AKI) during their hospital stay will participate in the ACT program which provides standardized education and assists with coordination of follow up care after hospital stay.
  Interventions: Behavioral: AKI in Care Transitions (ACT) program
- Usual Care Group (No Intervention): Subjects diagnosed with Acute Kidney Injury (AKI) during their hospital stay will receive standard of care from their inpatient and outpatient care teams.

INTERVENTIONS:
Behavioral: AKI in Care Transitions (ACT) program — Multicomponent transitional support bundle that includes consultation from nurse educators before discharge to deliver kidney health education and coordination of appointments post-discharge.
  Arms: AKI in Care Transitions (ACT) Group

SUMMARY:
This research is being done to develop materials and processes that will help facilitate education and kidney care coordination for AKI survivors.

ELIGIBILITY:
Inclusion Criteria:

- Participants will be recruited from those identified by a developed electronic health record list of patients with stage III AKI (severe) during a hospitalization based on serum creatinine rise or urine output decline from Olmsted County.

Exclusion Criteria:

* Dementia.
* Non-English speaking.
* Expected to be dismissed to a skilled nursing facility or hospice at discharge.
* Expected to need dialysis at discharge.
* Primary Care Transitions Program enrollment.
* Transplant recipients within 100 days of transplant.
* Can only have one time enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Barreto, PharmD, RPh, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] May HP, Griffin JM, Herges JR, Kashani KB, Kattah AG, Mara KC, McCoy RG, Rule AD, Tinaglia AG, Barreto EF. Comprehensive Acute Kidney Injury Survivor Care: Protocol for the Randomized Acute Kidney Injury in Care Transitions Pilot Trial. JMIR Res Protoc. 2023 May 22;12:e48109. doi: 10.2196/48109. PMID 37213187

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were identified using an electronic health record (EHR)- embedded list of adults (≥18 years) hospitalized at Mayo Clinic in Rochester from January 2022 to July 2023 who met stage 3 AKI criteria based on serum creatinine rise or urine output decline during a hospitalization and had a local address.
  Candidate participants were approached within 48-72 hours of discharge to obtain written informed consent and randomized 1:1 to the ACT intervention or usual care.
Period: Overall Study
Arm/Group | AKI in Care Transitions (ACT) Group | Usual Care Group
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AKI in Care Transitions (ACT) Group | Usual Care Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [56 to 74] | 66 [58 to 70] | 65 [56 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 17 | 18 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic Caucasian | 23 | 20 | 43
  Race/Ethnicity: Other or Unknown Race/Ethnicity | 2 | 5 | 7
Preadmission baseline eGFR [Median (Inter-Quartile Range); unit: mL/min/1.73m^2] | 63 [34 to 92] | 61 [43 to 69] | 62 [35 to 71]
Discharge eGFR [Median (Inter-Quartile Range); unit: mL/min/1.73m^2] | 31 [23 to 79] | 27 [20 to 50] | 30 [21 to 74]
AKI Recovery stage at discharge [Count of Participants; unit: Participants]
  Recovered (back to baseline) or stage 0 recovery (serum creatinine < 1.5x baseline) | 17 | 13 | 30
  Stage 1 recovery (1.5-1.9x baseline) | 3 | 5 | 8
  Stage 2 recovery (2.0-2.9x baseline) | 3 | 3 | 6
  Stage 3 recovery (3x baseline or >= 4 mg/dL) | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects to Complete the ACT Program
Description: Total number of subjects to complete the full ACT program intervention
Time Frame: 30 days after hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | AKI in Care Transitions (ACT) Group
Number analyzed (Participants) | 25
Participants | 22

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | AKI in Care Transitions (ACT) Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 1/25 | 1/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT05184894/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT05184894/ICF_000.pdf